CLINICAL TRIAL: NCT03188159
Title: Phase II Study of Intravenous Vinorelbine in Patients With Relapsed Platinum Resistant or Refractory C5 High Grade Serous, Endometrioid, or Undifferentiated Primary Peritoneum, Fallopian Tube or Ovarian Cancer (VIP)
Brief Title: Vinorelbine in Relapsed Platinum Resistant or Refractory C5 High Grade Serous, Endometrioid, or Undifferentiated Primary Peritoneum, Fallopian Tube or Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Cancer Centre, Singapore (Other); KK Women's and Children's Hospital (Other Government); Australia New Zealand Gynaecological Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GY01/05/16
Record Dates: First submitted 2017-03-16; First posted 2017-06-15 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV Vinorelbine (Experimental): IV Vinorelbine 25mg/m2
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine 25 mg/m2 intravenously on day-1 and day-8 of a 3 week cycle to commence following confirmation of eligibility into the study for a maximum of 12 months, until disease progression, intolerable toxicity or withdrawal of patient consent (whichever event occurs first).

SUMMARY:
This is a phase II study in patients with recurrent platinum resistant or refractory C5 high-grade serous, endometrioid or undifferentiated ovarian, primary peritoneal or fallopian tube cancer. All patients with high-grade serous, endometrioid or undifferentiated primary peritoneum, fallopian tube or ovarian cancer will be eligible to be screened for this trial and will be required to sign a pre-screening consent form.

DETAILED DESCRIPTION:
Background Therapeutic Information In ovarian cancer, several single agent phase II trials of vinorelbine in recurrent OC have shown variable response rates of 3 - 30%. However, previous studies have involved "all-comers" and no reported trials have selected patients based on confirmed pure HGSOC or a biomarker of relevance. Preclinical studies suggest that genes involved in microtubule dynamics, are significantly over-expressed in C5 tumours. Importantly, increased sensitivity was demonstrated of C5-like cell lines to tubulin depolymerising agents like vincristine and vinorelbine compared with microtubule stabilizing agents like paclitaxel. Subsequent studies on patient derived xenograft (PDX) models of C5 HGSOC (including platinum resistant models) showed responses for more than 50 days when treated with vinorelbine, providing preclinical proof that vinorelbine may be an effective therapeutic option in targeting the C5 subclass of HGSOC, including in platinum resistant or refractory disease.

Risk/ Benefit of Intervention Vinorelbine is a hemisynthetic vinca alkaloid that is traditionally administered intravenously via an infusion. The mechanism of action is disruption of microtubules by their reversible binding to tubulin resulting in mitotic spindle dissolution and metaphase arrest in dividing cells. This trial will afford patients with C5 relapsed platinum resistant or refractory HGSOC additional treatment options that may potentially have greater benefit than standard chemotherapy.

Tolerability The main dose limiting toxicity associated with IV vinorelbine in lung cancer is myelosuppression with Grade 3-4 neutropenia seen in up to 46% of patients. However, the febrile neutropenia rate was low at <5%. Mild to moderate gastrointestinal toxicity was observed with nausea and vomiting being the most common adverse effect. Grade 3/4 nausea or vomiting occurred in 7% - 17% of patients and primary prophylaxis is recommended. Neurotoxicity was also reported with the use of vinorelbine. Peripheral neuropathy was observed in up to 11% of patients,and neuroconstipation was documented to affect up to 24% of patients, however most of these cases were mild, grade 1-2. A similar toxicity profile was observed in patients with platinum resistant ovarian cancer treated with vinorelbine. Leukopenia was the most common dose limiting toxicity followed by anemia, fatigue and nausea.

Aim and Objectives of the trial The purpose of this trial is to determine if targeting platinum resistant or refractory C5 high-grade serous, high grade endometrioid or undifferentiated ovarian, primary peritoneal and fallopian tube with vinorelbine can improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent
2. Patients must have platinum resistant or refractory HGSOC; defined as progressive disease by imaging ≤ 6 months from last date of most recent platinum-based therapy or rising CA-125 based on GCIG criteria
3. Have histological confirmation of high-grade serous or high-grade endometrioid or undifferentiated tumour of the primary peritoneum, fallopian tube cancer or ovary
4. Molecular subtyping by Nanostring technology must confirm C5 subtype on primary ovarian surgical sample or a biopsy of recurrent disease
5. Patients must not have received more than 3 prior chemotherapy regimens, which may include chemotherapy, biologics or other targeted therapies (this does not include maintenance treatment or hormonal therapy) for platinum resistant disease
6. Measurable disease by RECIST criteria (version 1.1).
7. At time of registration, if the patient has had previous treatment it must have been at least 28 days since major surgery or radiation therapy; 28 days from any other previous anti-cancer therapy including biologics; 14 days since hormone therapy. Patients must have recovered to ≤ grade 1 from their treatment-related events with the exception of alopecia.
8. Age ≥ 18 years of age (Age ≥ 21 years of age for Singapore sites)
9. Have clinically acceptable laboratory screening results within certain limits specified below:

   * AST and ALT ≤ 2.5 times upper limit of normal (ULN)
   * Total bilirubin ≤ ULN
   * Creatinine ≤ 1.5 x UL
   * Absolute neutrophil count ≥ 1500 cells/mm
   * Platelets ≥ 100,000/mm3
   * Hemoglobin ≥ 9.0 g/dl
10. Have an ECOG performance status of ≤ 2.
11. Women of child-producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication.
12. Have the ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
13. Able to tolerate IV medication.
14. Life expectancy greater than 6 months

Exclusion Criteria:

1. Women who are pregnant or nursing
2. Previous exposure to vinorelbine
3. Patients known to be hypersensitive to vinorelbine or any vinca alkaloids previously
4. Persistent toxicities (≥ Common Terminology Criteria for Adverse Event (CTCAE) v4.0 grade 1) caused by previous cancer therapy, excluding alopecia
5. Have active, acute, or chronic clinically significant infections or bleeding.
6. Have active angina pectoris, stroke, myocardial infarction, or any other pre-existing uncontrolled cardiovascular condition within the last 6 months.
7. Have additional uncontrolled serious medical or psychiatric illness.
8. Require therapeutic doses of anti-coagulation with warfarin or warfarin derivatives. However, treatment with low molecular weight heparin (LMWH) is allowed.
9. Known symptomatic CNS metastases. Treated brain metastatis that are stable for more than ≥4 weeks are allowed.
10. Psychiatric disorders that would hinder compliance with study protocol
11. History of other malignancies within the past 5 years except for curatively treated skin BCC or SCC or cervical carcinoma in situ. Patients who have had curatively treated breast cancer, with completion of adjuvant chemotherapy more than three years before are allowed.
12. Require treatment with drugs known to be potent inducers or inhibitors of CYP3A4 at the time of registration
13. Subjects known to be HIV positive or with active and untreated Hepatitis B or Hepatitis C infection. Patients with controlled Hepatitis B or Hepatitis C infection on treatment with antiviral medication are allowed.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The disease is only contracted by females who have the organs (fallopian tube and ovaries).
Enrollment: 36 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Response rates | 3 years
  To determine the activity of vinorelbine as defined by response rates when patients with recurrent platinum resistant or refractory C5 high-grade serous, endometrioid or undifferentiated ovarian, primary peritoneal or fallopian tube cancer are treated with IV vinorelbine based on RECISTv1.1

SECONDARY OUTCOMES:
Progression free survival | 3 years
  To assess progression free survival when patients with recurrent platinum resistant C5 high-grade serous, endometrioid or undifferentiated ovarian, primary peritoneal and fallopian tube cancer are treated with IV vinorelbine
Changes in the level of CA 125 | 3 years
  A response according to CA 125 has occurred if there is at least a 50% reduction in CA 125 levels from a pretreatment sample. The response must be confirmed and maintained for at least 28 days. Patients can be evaluated according to CA 125 only if they have a pretreatment sample that is at least twice the upper limit of normal and within 2 weeks prior to starting treatment
Adverse event profile | 3 years
  To assess the adverse event profile of IV vinorelbine in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: David Tan, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Peter MacCallum Cancer Centre, Melbourne, Australia
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaughan S, Coward JI, Bast RC Jr, Berchuck A, Berek JS, Brenton JD, Coukos G, Crum CC, Drapkin R, Etemadmoghadam D, Friedlander M, Gabra H, Kaye SB, Lord CJ, Lengyel E, Levine DA, McNeish IA, Menon U, Mills GB, Nephew KP, Oza AM, Sood AK, Stronach EA, Walczak H, Bowtell DD, Balkwill FR. Rethinking ovarian cancer: recommendations for improving outcomes. Nat Rev Cancer. 2011 Sep 23;11(10):719-25. doi: 10.1038/nrc3144. PMID 21941283
- [Background] McGuire WP, Hoskins WJ, Brady MF, Kucera PR, Partridge EE, Look KY, Clarke-Pearson DL, Davidson M. Cyclophosphamide and cisplatin compared with paclitaxel and cisplatin in patients with stage III and stage IV ovarian cancer. N Engl J Med. 1996 Jan 4;334(1):1-6. doi: 10.1056/NEJM199601043340101. PMID 7494563
- [Background] ICON2: randomised trial of single-agent carboplatin against three-drug combination of CAP (cyclophosphamide, doxorubicin, and cisplatin) in women with ovarian cancer. ICON Collaborators. International Collaborative Ovarian Neoplasm Study. Lancet. 1998 Nov 14;352(9140):1571-6. PMID 9843101
- [Background] Ozols RF, Bundy BN, Greer BE, Fowler JM, Clarke-Pearson D, Burger RA, Mannel RS, DeGeest K, Hartenbach EM, Baergen R; Gynecologic Oncology Group. Phase III trial of carboplatin and paclitaxel compared with cisplatin and paclitaxel in patients with optimally resected stage III ovarian cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2003 Sep 1;21(17):3194-200. doi: 10.1200/JCO.2003.02.153. Epub 2003 Jul 14. PMID 12860964